CLINICAL TRIAL: NCT01143402
Title: Randomized Phase II Trial of Temozolomide Versus Hyd-Sulfate AZD6244 [NSC 748727] in Patients With Metastatic Uveal Melanoma
Brief Title: Temozolomide or Selumetinib in Treating Patients With Metastatic Melanoma of the Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01411; NCI-2011-01411 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000674866; 10-053 (Other: Memorial Sloan-Kettering Cancer Center); 8443 (Other: CTEP); N01CM00070 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); N01CM00100 (NIH); N01CM62206 (NIH); N01CM62208 (NIH); P30CA008748 (NIH); U01CA132123 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Iris Melanoma; Medium/Large Size Posterior Uveal Melanoma; Ocular Melanoma With Extraocular Extension; Recurrent Uveal Melanoma; Small Size Posterior Uveal Melanoma; Stage IV Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Dacarbazine; AZD 6244; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who are unable to be treated with temozolomide may be treated with dacarbazine IV every 3 weeks (with approval from the Principal Investigator). Patients who experience disease progression may crossover to arm II.
  Interventions: Drug: Dacarbazine; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Temozolomide
- Arm II (selumetinib) (Experimental): Patients receive selumetinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Selumetinib

INTERVENTIONS:
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
  Arms: Arm I (temozolomide)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244
  Arms: Arm II (selumetinib)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac
  Arms: Arm I (temozolomide)

SUMMARY:
This randomized phase II trial studies temozolomide to see how well it works compared to selumetinib in treating patients with melanoma of the eye that has spread to other places in the body. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether temozolomide is more effective than selumetinib in treating melanoma of the eye.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the progression-free survival (PFS) in three separate patient populations with uveal melanoma: Patients on COHORT 1 (guanine nucleotide binding protein [G protein], q polypeptide [Gnaq]/G protein, alpha 11 [Gna11] mutant uveal melanoma; temozolomide [TMZ]/dacarbazine [DTIC] naive) treated with AZD6244 (selumetinib) or TMZ (or DTIC); patients on both COHORT 1 and COHORT 2 (Gnaq/Gna11 mutant and Gnaq/Gna11 wild-type uveal melanoma; TMZ/DTIC naive) treated with AZD6244 or TMZ (or DTIC); and patients on COHORT 3 (Gnaq/Gna11 mutant or wild-type uveal melanoma; previously treated with TMZ/DTIC) treated with AZD6244.

SECONDARY OBJECTIVES:

I. Overall survival (OS). II. Overall response rate (RR). III. To determine the tolerability of AZD6244 in patients with advanced uveal melanoma.

IV. To correlate PFS, OS, and overall RR with Gnaq and Gna11 mutational status.

TERTIARY OBJECTIVES:

I. To correlate clinical outcome with baseline phosphorylated (p)-extracellular signal-regulated kinases (ERK), p-v-akt murine thymoma viral oncogene homolog 1 (AKT), and phosphatase and tensin homolog (PTEN) expression by immunohistochemistry.

II. To correlate clinical outcome with changes in p-ERK, p-AKT, and PTEN expression by immunohistochemistry.

III. To correlate clinical outcome with changes in Ki67 and cleaved caspase 3. IV. To explore the overall quality of life (QoL) of the treatment groups as measured by the Functional Assessment of Cancer Therapy-Melanoma (FACT-M) questionnaire.

V. To explore the radiographic effects of treatment with AZD6244 as assessed by 18F fluorothymidine (FLT)-positron emission tomography (PET) imaging.

OUTLINE: Patients in groups 1 and 2 are randomized to 1 of 2 treatment arms. Patients in group 3 are assigned to arm II.

ARM I: Patients receive temozolomide orally (PO) once daily (QD) on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who are unable to be treated with temozolomide may be treated with dacarbazine intravenously (IV) every 3 weeks (with approval from the Principal Investigator). Patients who experience disease progression may crossover to arm II.

ARM II: Patients receive selumetinib PO twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic histologically or cytologically confirmed uveal melanoma; if histologic or cytologic confirmation of the primary is not available, confirmation of the primary diagnosis of uveal melanoma by the treating investigator can be clinically obtained, as per standard practice for uveal melanoma; pathologic confirmation of diagnosis will be performed at Memorial Sloan-Kettering Cancer Center (MSKCC) or at a participating site
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL (not requiring transfusions within the past 2 weeks)
* Total bilirubin =< 1.5 times upper limit of normal; note: patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times upper limit of normal for patients with no concurrent liver metastases
* AST(SGOT)/ALT(SGPT) =< 5 X institutional ULN for patients with concurrent liver metastases
* Creatinine =< 1.5 mg/dL
* Tumor Gnaq and Gna11 status must be determined on all patients using a Clinical Laboratory Improvement Act (CLIA) approved assay; if initial CLIA testing is performed locally, patients must consent to provide a tumor block or unstained slides to MSKCC for central review of Gnaq and Gna11 status; this central review may be performed retrospectively and will not delay patient treatment on study
* Patients must agree to provide all imaging studies for central radiology review; this central radiology review may be performed retrospectively and will not be utilized for decision making for patients on study
* Ability to understand and the willingness to sign a written informed consent document
* Eligibility for enrollment in each cohort is dependent upon tumor Gnaq/Gna11 status and prior therapy as follows:

  * Cohort 1: no prior TMZ or DTIC; mutant Gnaq/Gna11 status
  * Cohort 2: no prior TMZ or DTIC; wild-type Gnaq/Gna11 status
  * Cohort 3: received prior TMZ or DTIC; mutant or wild-type Gnaq/Gna11 status
* Every effort must be made to avoid administration of drugs that are inhibitors or inducers of cytochrome P450 1A2 (CYP1A2) and CYP3A4

Exclusion Criteria:

* Patients may have had any number of prior therapies, but cannot have previously been treated with a mitogen-activated protein kinase kinase (MEK) inhibitor; at least 3 weeks must have elapsed since the last dose of systemic therapy; at least 6 weeks must have elapsed if the last regimen included carmustine (BCNU), mitomycin C or an anti-CTLA4 antibody; patients must have experienced disease progression on their prior therapy in the opinion of the treating investigator
* Patients may not be receiving any other investigational agents
* Patients with active or untreated brain metastases; treated brain metastases must have been stable for at least 2 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TMZ or DTIC or AZD6244
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or bleeding, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breast-feeding should be discontinued if the mother is treated with AZD6244
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of child-bearing potential must have a negative pregnancy test prior to entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; please note that the AZD6244 manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; patients with compensated HIV, with adequate cluster of differentiation (CD)4+ T-cell counts, and not requiring antiretroviral medication will be allowed
* Patients taking vitamin E supplements while on study
* No concomitant anti-cancer chemotherapy or other systemic drugs; palliative radiation therapy will be allowed as long as the patient meets all other eligibility criteria
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Patients with corrected QT (QTc) interval > 450 msecs or other factors that increase the risk of QTc prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class III and IV definitions are excluded
* Every effort must be made to avoid the use of a concomitant medication that can prolong the QTc interval while receiving AZD6244; if the patient cannot discontinue medications that prolong the QTc interval while receiving AZD6244, close cardiac monitoring should be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (33):
- United States (32):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Wisconsin Clinical Cancer Center, Milwaukee, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Atkinson TM, Hay JL, Shoushtari A, Li Y, Paucar DJ, Smith SC, Kudchadkar RR, Doyle A, Sosman JA, Quevedo JF, Milhem MM, Joshua AM, Linette GP, Gajewski TF, Lutzky J, Lawson DH, Lao CD, Flynn PJ, Albertini MR, Sato T, Lewis K, Marr B, Abramson DH, Dickson MA, Schwartz GK, Carvajal RD. Relationship between physician-adjudicated adverse events and patient-reported health-related quality of life in a phase II clinical trial (NCT01143402) of patients with metastatic uveal melanoma. J Cancer Res Clin Oncol. 2017 Mar;143(3):439-445. doi: 10.1007/s00432-016-2318-x. Epub 2016 Dec 5. PMID 27921276
- [Derived] Carvajal RD, Sosman JA, Quevedo JF, Milhem MM, Joshua AM, Kudchadkar RR, Linette GP, Gajewski TF, Lutzky J, Lawson DH, Lao CD, Flynn PJ, Albertini MR, Sato T, Lewis K, Doyle A, Ancell K, Panageas KS, Bluth M, Hedvat C, Erinjeri J, Ambrosini G, Marr B, Abramson DH, Dickson MA, Wolchok JD, Chapman PB, Schwartz GK. Effect of selumetinib vs chemotherapy on progression-free survival in uveal melanoma: a randomized clinical trial. JAMA. 2014 Jun 18;311(23):2397-405. doi: 10.1001/jama.2014.6096. PMID 24938562
- [Derived] Chen X, Schwartz GK, DeAngelis LM, Kaley T, Carvajal RD. Dropped head syndrome: report of three cases during treatment with a MEK inhibitor. Neurology. 2012 Oct 30;79(18):1929-31. doi: 10.1212/WNL.0b013e318271f87e. Epub 2012 Oct 17. No abstract available. PMID 23077008

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Temozolomide): Randomized to Temozolomide
- Arm II (Selumetinib): Randomized to Selumetinib
- Non-Randomized (Selumetinib): Non-Randomized to Selumetinib
Period: Overall Study
Arm/Group | Arm I (Temozolomide) | Arm II (Selumetinib) | Non-Randomized (Selumetinib)
Started | 51 | 50 | 19
Completed | 50 | 49 | 18
Not Completed | 1 | 1 | 1
Not completed — Rapid clinical decline | 1 | 1 | 0
Not completed — Not Treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Temozolomide) | Arm II (Selumetinib) | Non-Randomized (Selumetinib) | Total
Number analyzed (Participants) | 51 | 50 | 19 | 120
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 86] | 62 [32 to 86] | 63 [42 to 81] | 62 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 10 | 54
  Male | 31 | 26 | 9 | 66

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Evaluable Randomized Patients)
Description: The primary analysis will be performed among the Gnaq/Gna11 mutant patients. A stratified logrank test will be performed stratified by mutation status, M stage, and number of prior systemic therapies for metastatic disease. Due to the potential for a large number of strata and small strata sizes, the standard asymptotic stratified logrank test will be verified for robustness utilizing a permutation reference distribution.
Time Frame: The time from randomization to the earlier date of objective disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) criteria or death due to any cause in the absence of progression, assessed up to 5 years
Population: Analysis of progression-free survival in all evaluable randomized patients
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm I (Temozolomide) | Arm II (Selumetinib)
Number analyzed (Participants) | 49 | 47
weeks | 7 [4.3 to 8.4] | 15.9 [8.4 to 21.1]

2. Secondary Outcome: Median Overall Survival (Evaluable Randomized Patients)
Description: as for outcome 1
Time Frame: The time from randomization to death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Temozolomide) | Arm II (Selumetinib)
Number analyzed (Participants) | 50 | 49
Months | 9.1 [6.1 to 11.1] | 11.8 [9.8 to 15.7]

3. Other Pre Specified Outcome: Objective Disease Progression
Description: per Response Evaluation Criteria In Solid Tumors (RECIST) criteria or death due to any cause in the absence of progression
Time Frame: assessed up to 5 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Survival
Description: as for outcome 1
Time Frame: The time from randomization to death due to any cause, assessed up to 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Response Rate (Complete and Partial Response)
Description: Calculated along with a 95% confidence interval.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Toxicity According to the National Cancer Institute Common Toxicity Criteria
Description: Toxicity will be reported by type, frequency, and severity. Please see adverse events.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PFS (Group 3)
Description: Evaluated using a Simon mini-max design. Curves will be generated using Kaplan-Meier methodology.
Time Frame: 4 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Apoptosis in the Paired Samples, Performed by Caspase 3 Cleavage
Description: Changes will be assessed by a Wilcoxon test
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Ki67
Description: Correlated with disease status using Fishers exact test.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in p-AKT
Description: Correlated with disease status using Fishers exact test.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in p-ERK
Description: Decrease in p-ERK will be correlated with disease status using Fishers exact test.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in PTEN
Description: Correlated with disease status using Fishers exact test.
Time Frame: Baseline up to 4 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in Maximum Standardized Uptake Value on FLT-PET Scans
Description: A paired student's t-test will be performed. Analysis of variance will also be performed to obtain the significance of FLT-PET uptake on each lesion between patients.
Time Frame: Baseline up to 60 minutes post injection
Reporting Status: Not Posted

14. Other Pre Specified Outcome: FACT-M Total Score
Description: Summarized using descriptive statistics for each assessment time and by treatment group. The scores will be compared between treatment groups using a mixed effect model for repeated measures analysis method. Treatment difference will be estimated from the model for each assessment time.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm I (Temozolomide) | Arm II (Selumetinib) | Non-Randomized (Selumetinib)
Serious Adverse Events (participants affected / at risk) | 18/50 | 19/49 | 7/18
Other Adverse Events (participants affected / at risk) | 50/50 | 49/49 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Temozolomide) (N=50) | Arm II (Selumetinib) (N=49) | Non-Randomized (Selumetinib) (N=18)
Abdominal pain (General disorders) | 1 | 2 | 0
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1 | 2 | 1
Ascites (General disorders) | 1 | 0 | 0
CPK increased (Blood and lymphatic system disorders) | 4 | 9 | 2
Creatinine increased (Metabolism and nutrition disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Neoplasms (Skin and subcutaneous tissue disorders) | 9 | 3 | 4
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 0 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Thromboembolic event (Cardiac disorders) | 1 | 1 | 0
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 0 | 2 | 0
Blood bilirubin increased (Metabolism and nutrition disorders) | 0 | 3 | 1
Confusion (General disorders) | 0 | 1 | 0
Death NOS (General disorders) | 0 | 1 | 0
Dehydration (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Edema limbs (General disorders) | 0 | 1 | 0
GGT increased (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nausea (Blood and lymphatic system disorders) | 0 | 1 | 0
Syncope (General disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
General Disorders (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Temozolomide) (N=50) | Arm II (Selumetinib) (N=49) | Non-Randomized (Selumetinib) (N=18)
Anemia (Blood and lymphatic system disorders) | 8 | 15 | 6
Leukopenia (Blood and lymphatic system disorders) | 9 | 6 | 6
Lymphopenia (Blood and lymphatic system disorders) | 5 | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5 | 5
Alanine Amino Transferase Elevation (Blood and lymphatic system disorders) | 4 | 21 | 7
Alopecia (General disorders) | 0 | 6 | 1
Anorexia (General disorders) | 7 | 4 | 1
Arthralgias (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Aspartate Amino Transferase Elevation (Blood and lymphatic system disorders) | 6 | 25 | 7
Blurred Vision (Eye disorders) | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 15 | 3 | 1
CPK Elevation (General disorders) | 0 | 26 | 14
Diarrhea (Gastrointestinal disorders) | 4 | 20 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 2
Edema Face (General disorders) | 0 | 6 | 3
Eye Disorder (Eye disorders) | 0 | 4 | 1
Fatigue (General disorders) | 22 | 30 | 8
Mucositis (General disorders) | 1 | 6 | 0
Nausea (Gastrointestinal disorders) | 20 | 18 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 8 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 3 | 38 | 12
Vomiting (Gastrointestinal disorders) | 12 | 11 | 3
Edema Limbs (General disorders) | 1 | 15 | 10

LIMITATIONS AND CAVEATS:
Limitations of this study include the unblinded trial design and the lack of central review of imaging studies. Additionally, this trial was designed before activating mutations in exon 4 of GNAQ and GNA11 were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less